CLINICAL TRIAL: NCT01783418
Title: A Randomized, Wait-list Controlled Clinical Trial: the Effects of a Mindfulness-based Intervention on Quality of Life, Sleep and Mood in Adolescents With Cancer.
Brief Title: Mindfulness-based Intervention for Teenagers With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Catherine Malboeuf-Hurtubise, Ph.D. Candidate, clinical psychology, Université de Montréal, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3550
Record Dates: First submitted 2013-01-29; First posted 2013-02-04 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Pediatric Cancer
Keywords: mindfulness-based meditation; pediatric cancer; adolescence; quality of life; sleep; affect; health psychology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness intervention (Experimental)
  Interventions: Behavioral: Mindfulness Intervention
- Wait-list control (Active Comparator)
  Interventions: Behavioral: Mindfulness Intervention

INTERVENTIONS:
Behavioral: Mindfulness Intervention — Mindfulness-based intervention adapted for teenagers

SUMMARY:
The purpose of this study is to evaluate the effects of a mindfulness-based meditation intervention on quality of life, sleep and mood in adolescents with cancer compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers (ages 12-18) with cancer

Exclusion Criteria:

* No ongoing or lifetime severe psychopathology, such as schizophrenia, psychosis, delusional disorders or organic mental disorders

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Malboeuf-Hurtubise, Ph.D. candidate, Principal Investigator — Université de Montréal; Marie Achille, Ph.D., Study Director — Université de Montréal; Serge Sultan, Ph.D., Study Director — Université de Montréal, St. Justine's Hospital; Majorie Vadnais, M.D., Study Director — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Mother and Child University Hospital Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Malboeuf-Hurtubise C, Achille M, Sultan S, Vadnais M. Mindfulness-based intervention for teenagers with cancer: study protocol for a randomized controlled trial. Trials. 2013 May 10;14:135. doi: 10.1186/1745-6215-14-135. PMID 23663534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the experimental condition, over 9 months of recruitment, 481 youth were screened for participation in this project. Of these, 418 were excluded. Of the 63 remaining, only 13 agreed to participate, gave their consent, and provided a complete dataset.
Pre-assignment Details: Over 9 months of recruitment, 481 youth were screened for participation in this project. Of these, 418 (86.9%) were excluded because they lived further than 1 hour from the intervention site, had no history of cancer, had died or were not reachable by telephone. Recruitment for the control group was completed shortly after.
Groups:
- No Treatment Control: Mindfulness Intervention: Mindfulness-based intervention adapted for teenagers
Period: Overall Study
Arm/Group | Mindfulness Intervention | No Treatment Control
Started | 8 | 6
Completed | 7 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Intervention | No Treatment Control | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (0.9) | 15.3 (2.2) | 15.4 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mood From Baseline to Post-intervention and 6 Months Post-intervention
Description: Beck Youth Inventory - Anxiety scale Subscale range: 0 (minimum score) - 60 (maximum score)
  Higher scores indicate higher anxiety and a worse outcome
Time Frame: Baseline, Post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Intervention | No Treatment Control
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 18.9 (8.6) | 17.8 (6.9)
  Post-intervention (8 weeks) | 15.9 (6.7) | 12.8 (3.2)
Statistical Analysis 1: Comparison: Mindfulness Intervention vs No Treatment Control; Baseline and Post-intervention (8 weeks); Test type: Superiority or Other; p = 0.613, ANOVA

2. Primary Outcome: Changes in Quality of Life From Baseline to Post-intervention and 6 Months Post-intervention
Description: Pediatric Cancer Quality of Life Inventory
  Scale range: 0 (minimum score) to 108 (maximum score) Higher scores represent better outcomes
Time Frame: Baseline, Post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Intervention | No Treatment Control
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 73.8 (14.4) | 77.9 (10.3)
  Post-intervention (8 weeks) | 77.4 (11.8) | 81.6 (7.3)
Statistical Analysis 1: Comparison: Mindfulness Intervention vs No Treatment Control; Baseline, Post-intervention (8 weeks); Test type: Superiority or Other; p = 0.957, ANOVA

3. Primary Outcome: Changes Sleep From Baseline to Post-intervention and 6 Months Post-intervention
Description: Pittsburgh Sleep Quality Index
  Score range: 0 (minimum score) - 21 (maximum score)
  Higher scores indicate worse outcomes
Time Frame: Baseline, Post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Intervention | No Treatment Control
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 8.5 (4.6) | 6.5 (3.7)
  Post-intervention (8 weeks) | 6.5 (3.7) | 5.8 (2.8)
Statistical Analysis 1: Comparison: Mindfulness Intervention vs No Treatment Control; Baseline, Post-intervention (8 weeks); Test type: Superiority or Other; p = .256, ANOVA

4. Secondary Outcome: Changes in Mindfulness Propensity and Skills From Baseline to Post-intervention and 6 Months Post-intervention
Description: Children and Adolescent Mindfulness Measure Score range: 0 (minimum score) - 40 (maximum score)
  Higher scores represent better outcomes
Time Frame: Baseline, Post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Intervention | No Treatment Control
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 24.1 (5.6) | 27.8 (4.7)
  Post-intervention (8 weeks) | 27.3 (7.3) | 27.8 (4.7)
Statistical Analysis 1: Comparison: Mindfulness Intervention vs No Treatment Control; Baseline, Post-intervention (8 weeks); Test type: Superiority or Other; p = 0.97, ANOVA

5. Primary Outcome: Changes in Mood From Baseline to Post-intervention and 6 Months Post-intervention
Description: Beck youth inventories - Depression scale
  Subscale range: 0 (minimum score) - 60 (maximum score)
  Higher scores a worse outcome
Time Frame: baseline, Post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Intervention | No Treatment Control
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 15.8 (9.1) | 10.3 (5.6)
  Post-intervention (8 weeks) | 9.8 (5.2) | 9.2 (4.7)
Statistical Analysis 1: Comparison: Mindfulness Intervention vs No Treatment Control; Baseline, Post-intervention; Test type: Superiority or Other; p = 0.241, ANOVA

6. Primary Outcome: Changes in Mood From Baseline to Post-intervention and 6 Months Post-intervention
Description: PANAS-C - Positive affect
  Score range: 0 (minimum score) - 50 (maximum score)
  High scores represent better outcomes
Time Frame: baseline, Post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Intervention | No Treatment Control
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 27.4 (6.8) | 28.3 (4.5)
  Post-intervention (8 weeks) | 29.7 (7.9) | 27.0 (3.4)
Statistical Analysis 1: Comparison: Mindfulness Intervention vs No Treatment Control; Baseline, Post-intervention (8 weeks); Test type: Superiority or Other; p = 0.358, ANOVA

7. Primary Outcome: Changes in Mood From Baseline to Post-intervention and 6 Months Post-intervention
Description: PANAS-C - Negative affect
  Score range: 0 (minimum score) - 50 (maximum score) Higher scores represent worse outcomes
Time Frame: Baseline, Post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Intervention | No Treatment Control
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 19.7 (8.4) | 19.0 (4.0)
  Post-intervention (8 weeks) | 16.9 (4.5) | 16.3 (5.8)
Statistical Analysis 1: Comparison: Mindfulness Intervention vs No Treatment Control; Baseline, Post-intervention (8 weeks); Test type: Superiority or Other; p = 0.95, ANOVA

ADVERSE EVENTS:
Arm/Group | Mindfulness Intervention | No Treatment Control
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Major recruitment and retention issues leading to very small number of subjects recruited and analyzed.

Small sample leading to underpowered study and uninterpretable data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes